CLINICAL TRIAL: NCT00551733
Title: Paclitaxel Poliglumex (CT-2103)/Carboplatin vs Paclitaxel/Carboplatin for the Treatment of Chemotherapy-Naïve Advanced Non-Small Cell Lung Cancer (NSCLC) in Women With Estradiol >30 pg/mL
Brief Title: Carboplatin With Either Paclitaxel Poliglumex or Paclitaxel in Treating Women With Stage IIIB, Stage IV, or Recurrent Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CTI-PGT-07-00400; CDR0000573340 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2007-004167-22
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel; paclitaxel poliglumex

ARMS (2):
- Arm I (Experimental): Patients receive paclitaxel poliglumex IV over 10 minutes followed by carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: carboplatin; Drug: paclitaxel poliglumex
- Arm II (Active Comparator): Patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: carboplatin — Given IV
Drug: paclitaxel — Given IV
  Arms: Arm II
Drug: paclitaxel poliglumex — Given IV
  Arms: Arm I

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin, paclitaxel, and paclitaxel poliglumex, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving carboplatin together with paclitaxel poliglumex is more effective than giving carboplatin together with paclitaxel in treating non-small cell lung cancer.

PURPOSE: This randomized phase III trial is studying carboplatin and paclitaxel poliglumex to see how well they work compared with carboplatin and paclitaxel in treating women with stage III, stage IV, or recurrent non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the overall survival of patients with chemotherapy-naïve stage IIIB or IV or recurrent non-small cell lung cancer treated with paclitaxel poliglumex and carboplatin vs paclitaxel and carboplatin.

Secondary

* Compare the progression-free survival of women treated with these regimens.
* Compare the disease control in women treated with these regimens.
* Compare the clinical benefit in women treated with these regimens.
* Compare the response rate in women treated with these regimens.
* Compare the quality of life of women treated with these regimens.
* Compare the safety and tolerability in women treated with these regimens.

OUTLINE: This is a multicenter study.

Patients are stratified according to age (≥ 60 vs < 60 years old), geographical location (United States of America, Canada, or Australia vs the rest of the world), extent of disease (independent of brain metastases, i.e., brain metastases are not considered in determining extent of disease) (intrathoracic disease only vs extrathoracic disease), and ECOG performance status (0 or 1 vs 2). Patients will be randomized to 1 of 2 treatment arms.

* Arm I: Patients receive paclitaxel poliglumex IV over 10 minutes followed by carboplatin IV over 30 minutes on day 1.
* Arm II: Patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes on day 1.

In both arms, treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, before each course, and at the completion of study treatment by the Pain Assessment Patient Questionnaire, the Pulmonary Symptom Index, and the Functional Assessment of Cancer Therapy- Lung Cancer Subscale (FACT-LCS) (only in countries in which a validated translation is currently available).

After completion of study therapy, patients are followed at least monthly.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed diagnosis of non-small cell lung cancer (NSCLC)

  * Cytologic specimens obtained by brushings, washings, or needle aspiration of a defined lesion or from a pleural effusion are acceptable; sputum cytology alone is not acceptable for determining cell type
* Must meet one of the following criteria:

  * Recurrent disease following completion of radiation or surgery
  * Stage IIIB disease and not a candidate for combined modality therapy (primary radiation therapy or surgery)
  * Stage IV disease
* Patients may have either measurable or nonmeasurable disease according to RECIST criteria
* Baseline estradiol > 30 pg/mL

  * Patients on hormone replacement therapy are eligible provided baseline estradiol > 30 pg/mL
* Patients with known brain metastases must have received standard antitumor treatment (e.g. whole brain radiation, stereotactic radioablation, or surgery) for their CNS metastases as defined by the site's institutional standards

  * Neurologic function must have been stable for 2 weeks before randomization and patients must either be off steroid therapy for their brain metastases or on a tapering regimen
  * Patients must have recovered from therapy for their brain metastases with no evidence of significant unstable neurological symptoms within the 4 weeks before study randomization
* No evidence of small cell carcinoma, carcinoid, or mixed small cell/non-small cell histology

PATIENT CHARACTERISTICS:

* Female
* ECOG performance score 0-2
* Life expectancy ≥ 12 weeks
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL (may be achieved with transfusion)
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 times ULN (CTC grade 1) (patients with Gilbert syndrome or other hereditary bilirubin defects may be included regardless of bilirubin levels)
* SGOT and SGPT ≤ 2.5 times ULN (CTC grade 0 or 1) (5 times ULN [CTC grade 0 to 2] if due to liver metastases)
* Alkaline phosphatase ≤ 2.5 times ULN except for elevated alkaline phosphatase with laboratory documentation that demonstrates bone origin
* No pregnant women or nursing mothers
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study participation
* No known hypersensitivity to study drugs or excipients
* Meets all of the following criteria:

  * No weight loss > 10% in previous 6 months
  * Lactate dehydrogenase (LDH) ≤ 600 IU/L (central laboratory) regardless of weight loss
  * LDH ≤ 400 IU/L (central laboratory) and no weight loss ≥ 5% in previous 6 months
  * BMI ≤ 35
* No concurrent primary malignancies except for carcinoma in situ or non-melanoma skin cancer
* No neuropathy grade 2 or greater
* No clinically significant active infection for which active therapy is underway
* No unstable medical conditions including unstable angina or myocardial infarction within the past 6 months

  * Patients with evidence of cardiac conduction abnormalities are eligible if their cardiac status is stable
* No circumstance that would preclude completion of the study or the required follow-up

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from major surgery
* At least 7 days since prior local palliative radiotherapy
* At least 30 days since prior radiation therapy with curative intent
* At least 4 weeks since prior investigational therapy, unless local requirements are more stringent
* No prior systemic chemotherapy for the treatment of lung cancer, including systemic radiosensitizers used to treat brain metastases or any biologic agents
* No concurrent non-protocol-specified systemic antitumor therapy
* No concurrent amifostine, investigational agents, other cytotoxic agents for this disease
* No concurrent radiotherapy (with the exception of radiotherapy for brain or bone metastases for palliative purposes or radiotherapy for a condition other than NSCLC that was ongoing at the time of randomization)

  * Patients receiving palliative radiotherapy (treatment for symptomatic metastatic disease) may be treated while on study

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2007-08 (Actual); Primary Completion 2007-12-25 (Actual); Study Completion 2007-12-25 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Progression-free survival
Disease control
Clinical benefit as defined by use of opiates, growth factors, and transfusions,
Response rate as assessed by complete response or partial response per RECIST criteria
Quality of life as assessed by Fact-LCS Scores and Pulmonary Symptom Index (PSI) Scores and Pain Scores
Safety as assessed by NCI CTCAE Version 3

CONTACTS AND LOCATIONS:
Overall Officials: Fred B. Oldham, MD, Study Chair — CTI BioPharma
Locations (41):
- United States (41):
  - Scottsdale Medical Specialists, Scottsdale, Arizona
  - Roy and Patricia Disney Family Cancer Center at Providence Saint Joseph Medical Center, Burbank, California
  - Southwest Cancer Care - Escondido, Escondido, California
  - Clinical Trials and Research Associates, Incorporated, Montebello, California
  - Stanford Cancer Center, Stanford, California
  - Broward Oncology Associates, Fort Lauderdale, Florida
  - Horizon Institute for Clinical Research, Hollywood, Florida
  - Rush Cancer Institute at Rush University Medical Center, Chicago, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Hematology Oncology Consultants - Naperville, Naperville, Illinois
  - Saint James Hospital and Health Centers Comprehensive Cancer Institute - Olympia Fields, Olympia Fields, Illinois
  - Cancer Center of Indiana, New Albany, Indiana
  - Providence Medical Group, Terre Haute, Indiana
  - Family Medicine of Vincennes Clinical Trial Center, Vincennes, Indiana
  - West Michigan Regional Cancer and Blood Center, Free Soil, Michigan
  - Newland Medical Associates PC - Southfield, Southfield, Michigan
  - Hattiesburg Clinic, PA at Forrest General, Hattiesburg, Mississippi
  - Columbia Comprehensive Cancer Care Clinic, Columbia, Missouri
  - Kansas City Cancer Centers - South, Kansas City, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Las Vegas Cancer Center, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Reno, Reno, Nevada
  - Richmond University Medical Center, Staten Island, New York
  - Lincoln Medical and Mental Health Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - Blood and Cancer Center, Incorporated, Canfield, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Vita Hematology Oncology at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Cancer Centers of the Carolinas - Eastside, Greenville, South Carolina
  - Family Cancer Center, PLLC - Collierville, Collierville, Tennessee
  - Mid-South Cancer Center, Germantown, Tennessee
  - Southwest Regional Cancer Center - Central, Austin, Texas
  - Lone Star Oncology - Austin, Austin, Texas
  - Mary Crowley Medical Research Center at Sammons Cancer Center, Dallas, Texas
  - Utah Hematology Oncology, PC, Ogden, Utah
  - Cancer Outreach Associates - Abingdon, Abingdon, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Cell Therapeutics, Incorporated, Seattle, Washington

REFERENCES:
- [Result] Langer CJ, O'Byrne KJ, Socinski MA, Mikhailov SM, Lesniewski-Kmak K, Smakal M, Ciuleanu TE, Orlov SV, Dediu M, Heigener D, Eisenfeld AJ, Sandalic L, Oldham FB, Singer JW, Ross HJ. Phase III trial comparing paclitaxel poliglumex (CT-2103, PPX) in combination with carboplatin versus standard paclitaxel and carboplatin in the treatment of PS 2 patients with chemotherapy-naive advanced non-small cell lung cancer. J Thorac Oncol. 2008 Jun;3(6):623-30. doi: 10.1097/JTO.0b013e3181753b4b. PMID 18520802